CLINICAL TRIAL: NCT06944041
Title: Limb Volumetry Using iPad Based 3D Scanner for Assessment of Edema
Brief Title: Measuring Volume Using a 3D Scanner and iPad to Grade the Swelling of Legs
Status: Completed | Type: Observational
Sponsor: The RANE Center for Venous and Lymphatic Diseases at St. Dominic's Hospital (Other)
Responsible Party: Principal Investigator, Dr. Seshadri Raju, Principal Investigator, The RANE Center for Venous and Lymphatic Diseases at St. Dominic's Hospital
Other Study IDs: 2024-008-St. Dom
Record Dates: First submitted 2025-04-14; First posted 2025-04-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Limb Volume; Measuring Edema
Keywords: Leg swelling; 3-D Volumetry; phlebolymphedema; CEAP Clinical Class 3; Limb plethysmography; lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Twenty limbs from ten healthy volunteers
  Interventions: Other: STO3 sensor (Structure Inc., Boulder, CO)

INTERVENTIONS:
Other: STO3 sensor (Structure Inc., Boulder, CO) — The advent of Apple iPad based 3D scanner opens a new avenue for measuring limb volume. The latest ambient light scanner model was utilized for the current study. 3D scanning technology has gained broad industrial use, including the manufacturing of high-precision tools. A commercially available software package was used for limb volumetry.

SUMMARY:
We used a new and easy-to-measure iPad 3D scanner to measure swelling in lower limbs because current technology is not easily available or affordable. We want to see how reliable the measurements are and what might affect how consistent they are.

DETAILED DESCRIPTION:
Twenty limbs from ten healthy volunteers were scanned using an iPad-based Structure Sensor and software. Initial scans followed standard manufacturer instructions, but high variance rendered data unsuitable for clinical use. To improve accuracy, a standardized scanning protocol was developed, incorporating anatomical calibration, scanning distance standardization, and scanning time control. A 254-mm calf segment was defined using a 3D marker placed on the medial malleolus to ensure consistent volume measurement. The scanning distance was fixed between 50-59 cm to reduce zoom parallax errors, and scans were conducted after 3 PM to minimize diurnal volume fluctuations. Multiple technicians performed repeat scans on the same limb to assess intra-observer and inter-observer scan reliability.

ELIGIBILITY:
Inclusion Criteria:

* The people in this study will be symptom free volunteers.

Exclusion Criteria:

* Pre-existing diseased limbs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population will be symptom-free volunteers in order to establish a method of scanning for the best results. Volunteers in this study will have no coercion involved.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Limb Volume | During Procedure
  The scanning protocol and the required modifications of "out of the box" instructions for optimal clinical application are described; The 10 inch (254mm) long limb segment scanned must be anatomically constant. We chose the medial malleolus as the lower border of the scan. The scannable limb volume is 254 mm long, measured up from the malleolus.

CONTACTS AND LOCATIONS:
Locations (1):
- The RANE Center for Venous and Lymphatic Diseases, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
The consent form clearly states that "We will not collect any protected health information in this study. Data collected will be as following: sex, age, weight, and volume of limbs." Therefore, there is no risk to patient confidentiality.

REFERENCES:
- [Background] Marsocci A, Santandrea S, Lanfranchi E, Donati D, Tedeschi R. Beyond water: 3D laser scanning offers a cutting-edge alternative for upper limb volume assessment. Phlebology. 2025 Jul;40(6):400-408. doi: 10.1177/02683555241310358. Epub 2024 Dec 19. PMID 39701043
- [Background] Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg. 2000 Jun;31(6):1307-12. doi: 10.1067/mva.2000.107094. PMID 10842165
- [Background] Raju S, Owen S Jr, Neglen P. Reversal of abnormal lymphoscintigraphy after placement of venous stents for correction of associated venous obstruction. J Vasc Surg. 2001 Nov;34(5):779-84. doi: 10.1067/mva.2001.119396. PMID 11700475
- [Background] Katz ML, Comerota AJ, Kerr RP, Caputo GC. Variability of venous-hemodynamics with daily activity. J Vasc Surg. 1994 Feb;19(2):361-5. doi: 10.1016/s0741-5214(94)70111-3. PMID 8114195